CLINICAL TRIAL: NCT02418130
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of 'Ursa Complex Soft Cap. (UDCA-004)' in Patients With Physical Fatigue.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_UDCA004
Record Dates: First submitted 2014-10-08; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Ursodeoxycholic Acid; Taurine; Ginsenosides; Thiamine; Inositol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- UDCA004 (Experimental): UDCA004
  Interventions: Drug: Ursodeoxycholic acid, taurine, ginsenoside, thiamine, inositol
- Placebo of UDCA004 (Placebo Comparator): Placebo of UDCA004
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursodeoxycholic acid, taurine, ginsenoside, thiamine, inositol
  Arms: UDCA004
Drug: Placebo
  Arms: Placebo of UDCA004

SUMMARY:
A multi-center, randomized, double-blind, placebo-controlled trial to evaluate the efficacy and safety of 'Ursa Complex Soft Cap. (UDCA-004)' in patients with physical fatigue.

ELIGIBILITY:
Inclusion Criteria:

* CIS greater than or equal to 76, HADS less than or equal to 10

Exclusion Criteria:

* Subjects who have diseases that can cause fatigue
* Subjects who are taking medication that can cause fatigue

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Rate of subjects whose CIS score has improved under 76 at week 4 | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seoul, South Korea